CLINICAL TRIAL: NCT05720416
Title: Effects of a Multi-intervention Programme on the Muscle Strength, Body Composition, Physical Performance and Quality of Life of the Elderly
Brief Title: Effects of a Multi-intervention Programme for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, assistant professor of nursing department, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202300020A3
Record Dates: First submitted 2022-09-07; First posted 2023-02-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Dementia
MeSH Terms: conditions — Sarcopenia; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- muscle strength training and protein supplementation (Experimental)
  Interventions: Dietary Supplement: protein supplementation; Behavioral: muscle strength training
- usual care (Placebo Comparator)
  Interventions: Other: usual care
- muscle strength training (Experimental)
  Interventions: Behavioral: muscle strength training

INTERVENTIONS:
Dietary Supplement: protein supplementation — protein supplementation for 16 weeks
  Arms: muscle strength training and protein supplementation
Behavioral: muscle strength training — muscle strength training for 16 weeks
  Arms: muscle strength training; muscle strength training and protein supplementation
Other: usual care — no intervention
  Arms: usual care

SUMMARY:
1. To develop a multiactivity training programme. 2. To explore the effect of this programme on sarcopenia, sarcopenic obesity, cognitive impairment and Parkinson's disease. 3. To compare the effects of the experimental and control treatments on the muscle strength, body composition, physical function performance and quality of life of the elderly.

ELIGIBILITY:
Inclusion Criteria:

(1) over 60 years old, (2) able to Communicate and follow instructions; (3) Stable condition with sufficient physical strength: able to maintain a seated position in a wheelchair or on the edge of a bed for at least one hour. (4) sarcopenia, sarcopenic obesity, cognitive impairment and Parkinson's disease.

Exclusion Criteria:

(1) difficulty in standing or walking and obvious musculoskeletal disease, (2) unsuitable for diagnosis by a physician those engaged in sports activities, (3) serious diseases/unstable states, such as severe heart, lung, liver and kidney diseases, severe malignant tumors, severe nutrition poor, severe dementia, (4) more than 180 minutes of exercise per week in the past month, (5) no willingness to participate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Chang in muscle strength from baseline to 16 weeks | Baseline and 16 weeks
  pinch, grip and quadriceps strength. A Higher score means a better outcome.
Chang in weight of muscle and fat from baseline to 16 weeks | Baseline and 16 weeks
  muscle mass(kg), fat mass (kg)
Chang in Activities of Daily Living from baseline to 16 weeks | Baseline and 16 weeks
  This is a scale of physical function. The range for total score is 0-100. A Higher score means a worse outcome.
Chang in Instrumental activities of daily living from baseline to 16 weeks | Baseline and 16 weeks
  This is a scale of physical function. The range for total score is 0-24. A Higher score means a better outcome.
Chang in Clinical Dementia Rating from baseline to 16 weeks | Baseline and 16 weeks
  Mental Function Assessment. The range is 0-3. A Higher score means a worse outcome.
Chang in Cornell Scale for Depression in Dementia from baseline to 16 weeks | Baseline and 16 weeks
  Mental Function Assessment. The range for total score is 0-38. A Higher score means a worse outcome.
Chang in Cohen-Mansfield Agitation Inventory from baseline to 16 weeks | Baseline and 16 weeks
  This is a scale of behavior measurement. The range for total is 29-203. A higher score means a worse outcome.
Chang in EQ5D from baseline to 16 weeks | Baseline and 16 weeks
  This is a scale of quality of life. The range for total is 0-20. A higher score means a worse outcome.
Chang in QUALIDEM from baseline to 16 weeks | Baseline and 16 weeks
  The scale is a dementia-specific Qol instrument. The range for total score is 0-120. A higher score means a better outcome.
Demographic attributes | Baseline
  Gender, education, age, married status, religion, medication, diseases, work and height.
Chang in PERSONAL WELLBEING INDEX from baseline to 16 weeks | Baseline and 16 weeks
  The range for total is 0-80. A higher score means a better outcome.
Chang in PERSONAL WELLBEING INDEX intellectual disability from baseline to 16 weeks | Baseline and 16 weeks.
  The range for total is 0-70. A higher score means a better outcome.
Chang in World Health Organization Quality of Life Instruments (WHOQOL-BREF) from baseline to 16 weeks | Baseline and 16 weeks.
  This is a scale of quality of life. The range for total is 26-130. A higher score means a better outcome.
Chang in Four-Meter Gait Speed from baseline to 16 weeks | Baseline and 16 weeks.
  Measured with seconds. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu, Principal Investigator — Central Taiwan University of Science and Technology
Locations (1):
- Daycare center at Central Taiwan University of Science and Technology, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No